CLINICAL TRIAL: NCT00913458
Title: A 3-Phase Study to Evaluate Sustained Remission and Productivity Outcomes in Subjects With Early Rheumatoid Arthritis Initiated on Treatment With Etanercept Plus Methotrexate
Brief Title: Study Evaluating Etanercept Plus Methotrexate in Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0881X1-4524; B1801020
Record Dates: First submitted 2009-05-26; First posted 2009-06-04 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Active Rheumatoid Arthritis; Arthritis, Rheumatoid; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): etanercept + methotrexate; etanercept + methotrexate
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept
  Other Names: Enbrel

SUMMARY:
Study to evaluate whether there is sustained remission and productivity in subjects with early rheumatoid arthritis started on etanercept plus methotrexate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early rheumatoid arthritis.
* Methotrexate (MTX) naive.
* Active early rheumatoid arthritis at the time of enrollment.

Exclusion Criteria:

* Previous or current treatment with etanercept, other tumor necrosis factor-alpha (TNF) inhibitors, or other biologic agents.
* Concurrent treatment with any disease-modifying anti-rheumatoid drugs (DMARD), within 4 weeks before baseline.
* Concurrent treatment with more than 1 non-steroidal anti-inflammatory drug (NSAID) at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- France (5):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
- Germany (11):
  - Pfizer Investigational Site, Vogelsang, Gommern
  - Pfizer Investigational Site, Altona
  - Pfizer Investigational Site, Elmshorn
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Ludwigsfelde
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Osnabrück
  - Pfizer Investigational Site, Rostock
  - Pfizer Investigational Site, Würzburg
  - Pfizer Investigational Site, Zerbst
- Pfizer Investigational Site, Dublin, Ireland, Ireland
- Italy (2):
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Pisa
- Pfizer Investigational Site, Monaco, Monaco
- Netherlands (3):
  - Pfizer Investigational Site, Amsterdam, North Holland
  - Pfizer Investigational Site, Haarlem
  - Pfizer Investigational Site, Heerlen
- Poland (8):
  - Pfizer Investigational Site, Ustroń, Poland
  - Pfizer Investigational Site, Warsaw, Poland
  - Pfizer Investigational Site, Żyrardów, Poland
  - Pfizer Investigational Site, Bydgoszczy
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, Doha, Qatar, Qatar
- Romania (3):
  - Pfizer Investigational Site, Bucharest, Romania
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Târgu Mureş
- Pfizer Investigational Site, Yaroslavl, Russia
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, A Coruña, La Coruna
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Barcelona, Spain
  - Pfizer Investigational Site, Valencia, Valencia
- Switzerland (3):
  - Pfizer Investigational Site, Sankt Gallen, Canton of St. Gallen
  - Pfizer Investigational Site, Chur
  - Pfizer Investigational Site, Lausanne
- United Kingdom (7):
  - Pfizer Investigational Site, Wigan, Lancaster
  - Pfizer Investigational Site, Manchester, Manchester
  - Pfizer Investigational Site, Harrogate, North Yorkshire
  - Pfizer Investigational Site, Dudley, West Midlands
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Tanaka Y, Smolen JS, Jones H, Szumski A, Marshall L, Emery P. The effect of deep or sustained remission on maintenance of remission after dose reduction or withdrawal of etanercept in patients with rheumatoid arthritis. Arthritis Res Ther. 2019 Jul 5;21(1):164. doi: 10.1186/s13075-019-1937-4. PMID 31277720
- [Derived] Fleischmann RM, van der Heijde D, Gardiner PV, Szumski A, Marshall L, Bananis E. DAS28-CRP and DAS28-ESR cut-offs for high disease activity in rheumatoid arthritis are not interchangeable. RMD Open. 2017 Jan 30;3(1):e000382. doi: 10.1136/rmdopen-2016-000382. eCollection 2017. PMID 28255449
- [Derived] Zhang W, Bansback N, Sun H, Pedersen R, Kotak S, Anis AH. Impact of etanercept tapering on work productivity in patients with early rheumatoid arthritis: results from the PRIZE study. RMD Open. 2016 Jul 7;2(2):e000222. doi: 10.1136/rmdopen-2015-000222. eCollection 2016. PMID 27486524
- [Derived] Wiland P, Dudler J, Veale D, Tahir H, Pedersen R, Bukowski J, Vlahos B, Williams T, Gaylord S, Kotak S. The Effect of Reduced or Withdrawn Etanercept-methotrexate Therapy on Patient-reported Outcomes in Patients with Early Rheumatoid Arthritis. J Rheumatol. 2016 Jul;43(7):1268-77. doi: 10.3899/jrheum.151179. Epub 2016 Jun 1. PMID 27252426
- [Derived] Zhang W, Bansback N, Sun H, Pedersen R, Kotak S, Anis AH. Estimating the monetary value of the annual productivity gained in patients with early rheumatoid arthritis receiving etanercept plus methotrexate: interim results from the PRIZE study. RMD Open. 2015 Apr 8;1(1):e000042. doi: 10.1136/rmdopen-2014-000042. eCollection 2015. PMID 26535135
- [Derived] Emery P, Hammoudeh M, FitzGerald O, Combe B, Martin-Mola E, Buch MH, Krogulec M, Williams T, Gaylord S, Pedersen R, Bukowski J, Vlahos B. Sustained remission with etanercept tapering in early rheumatoid arthritis. N Engl J Med. 2014 Nov 6;371(19):1781-92. doi: 10.1056/NEJMoa1316133. PMID 25372086
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4524&StudyName=Study%20Evaluating%20Etanercept%20plus%20Methotrexate%20in%20Early%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents the results of open-label 52-week treatment period (Phase 1), 39 week, double blind randomized (Phase 2) and 26 week observational period (Phase 3) part of a 121 week Phase 4 study program. Responders in Phase 1 were randomized to 3 arms (1:1:1 ratio) in Phase 2. Responders in Phase 2, continued to Phase 3 observational period
Pre-assignment Details: Phase 1 responders, defined as subjects with Disease Activity Score based on 28-joints count (DAS28) ≤ 3.2 at Week 39 and DAS28 <2.6 at Week 52, were randomized to Phase 2. The responders of Phase 2 were observed for 26-weeks in Phase 3 study that include 2 to 4 week period of double blind treatment taper of MTX followed by observational period
Groups:
- ETN 50 QW + MTX (Phase 1): Phase 1 was a 52-week open-label, single-arm period in which all subjects were treated with etanercept (ETN) 50 mg once weekly plus methotrexate (MTX). MTX starting dose was 10 mg per week and could increase by 5 mg per week increments up to Week 8, and up to a maximum of 25 mg per week. Participants with Disease Activity Score based on 28-joints count [DAS28] ≤3.2 at Week 39 and DAS28 <2.6 at Week 52 classified as a phase 1 responder, and will continue to Phase 2 study.
- E25 + MTX (Phase 2): In Phase 2 E25 + MTX arm, Etanercept 25 milligram (mg) was administered once weekly as a subcutaneous injection using the 25 mg pre filled syringe. Methotrexate was administered once weekly as oral capsules. All subjects received a dose of methotrexate during this Phase 2 study that was equal to their optimal methotrexate dose in earlier Phase 1 study. The subjects received the study treatment for 39 weeks, unless the subject was evaluated as non-responder at Week 64 or Week 76 and discontinued the study. Participants in sustained remission (Disease Activity Score based on 28-joints count [DAS28] <2.6) or with low disease activity (2.6 ≤ DAS28 ≤ 3.2) at Week 91 were classified as Phase 2 responder, and will continue to Phase 3 study.
- MTX + PBO (Phase 2): In Phase 2 MTX + PBO arm, the weekly dose of etanercept was tapered from the 50 mg dosage. At Week 52, subjects assigned to this arm received a double blinded 25 mg dose of etanercept as a subcutaneous injection using a pre filled syringe. All weekly doses thereafter (ie, Weeks 53 to 90) were administered as an etanercept matching placebo injection using a pre-filled syringe. Methotrexate was administered once weekly as oral capsules. All subjects received a dose of methotrexate during this Phase 2 study that was equal to their optimal methotrexate dose in earlier Phase 1 study. The subjects received the study treatment for 39 weeks, unless the subject was evaluated as non-responder at Week 64 or Week 76 and discontinued the study. Participants in sustained remission (Disease Activity Score based on 28-joints count [DAS28] <2.6) or with low disease activity (2.6 ≤ DAS28 ≤ 3.2) at Week 91 were classified as Phase 2 responder, and will continue to Phase 3 study.
- Placebo (PBO) (Phase 2): In Phase 2 Placebo (PBO) arm, the weekly dose of etanercept was tapered from the 50 mg dosage to a placebo injection. At Week 52, subjects assigned to this arm received a double blinded 25 mg dose of etanercept as a subcutaneous injection using a pre filled syringe. All weekly doses thereafter (ie, Weeks 53 to 90) were administered as an etanercept-matching placebo injection using a pre-filled syringe.
  Methotrexate-matching placebo was administered once weekly as oral capsules. The subjects received the study treatment for 39 weeks, unless the subject was evaluated as non-responder at Week 64 or Week 76 and discontinued the study. Participants in sustained remission (Disease Activity Score based on 28-joints count [DAS28] <2.6) or with low disease activity (2.6 ≤ DAS28 ≤ 3.2) at Week 91 were classified as Phase 2 responder, and will continue to Phase 3 study.
- E25+MTX (Phase 3); MTX (Phase 3); Placebo (PBO) (Phase 3): Phase 3 was a 26-week observational period in which Phase 2 responders progressively stopped treatment. It included a 2 to 4 week period of double blind MTX tapering (depending on the optimized MTX dose), followed by an observational period until Week 117.
Period: Phase 1
Arm/Group | ETN 50 QW + MTX (Phase 1) | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2) | E25+MTX (Phase 3) | MTX (Phase 3) | Placebo (PBO) (Phase 3)
Started | 306 | 0 (This arm is part of Phase 2 study) | 0 (This arm is part of Phase 2 study) | 0 (This arm is part of Phase 2 study) | 0 (This arm is part of Phase 3 study) | 0 (This arm is part of Phase 3 study) | 0 (This arm is part of Phase 3 study)
Completed | 194 (194 continued to Phase 2 but 1 was randomized in error leaving 193 in the phase 2 analysis.) | 0 (This arm is part of Phase 2 study) | 0 (This arm is part of Phase 2 study) | 0 (This arm is part of Phase 2 study) | 0 (This arm is part of Phase 3 study) | 0 (This arm is part of Phase 3 study) | 0 (This arm is part of Phase 3 study)
Not Completed | 112 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Responder | 54 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Request | 17 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 20 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 10 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Response per Investigator | 7 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | ETN 50 QW + MTX (Phase 1) | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2) | E25+MTX (Phase 3) | MTX (Phase 3) | Placebo (PBO) (Phase 3)
Started | 0 (This arm is part of Phase 1 of the study.) | 63 | 65 | 65 | 0 | 0 | 0
Completed | 0 (This arm is part of Phase 1 of the study.) | 53 (Participants randomized into Phase 3 of study.) | 46 (Participants randomized into Phase 3 of study.) | 32 (Participants randomized into Phase 3 of study.) | 0 | 0 | 0
Not Completed | 0 | 10 | 19 | 33 | 0 | 0 | 0
Not completed — Non-Responder | 0 | 5 | 7 | 12 | 0 | 0 | 0
Not completed — Subject Request | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Unsatisfactory Response per Investigator | 0 | 0 | 11 | 17 | 0 | 0 | 0
Period: Phase 3
Arm/Group | ETN 50 QW + MTX (Phase 1) | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2) | E25+MTX (Phase 3) | MTX (Phase 3) | Placebo (PBO) (Phase 3)
Started | 0 (This arm is part of Phase 1 of the study.) | 0 | 0 | 0 | 53 (Participants who completed Phase 2 study) | 46 (Participants who completed Phase 2 study) | 32 (Participants who completed Phase 2 study)
Completed | 0 (This arm is part of Phase 1 of the study.) | 0 | 0 | 0 | 31 | 28 | 24
Not Completed | 0 | 0 | 0 | 0 | 22 | 18 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Non-Responder | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Unsatisfactory Response per Investigator | 0 | 0 | 0 | 0 | 14 | 11 | 4

BASELINE CHARACTERISTICS:
Population: A total of 306 participants were enrolled in the study (Phase 1). Out of the 306 participants, 193 were eligible and were randomized at a ratio of 1:1:1 to Phase 2 study. Of the 193 participants from Phase 2, a total of 131 participants were eligible and were randomized to Phase 3 study.
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.94 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213
  Male | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Met Sustained Remission at Week 76 and Week 91 Based on DAS28 Score
Description: Sustained remission was defined as a DAS28 <2.6 at the Week 76 and Week 91 visits without requiring a corticosteroid boost between the Week 52 and Week 64 visits, where the requirement for a corticosteroid boost was defined as a value of DAS28 >3.2 at either the Week 56 or Week 64 visit.
  DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity.
  The participants who met sustained remission in both Week 76 and 91 are presented here.
Time Frame: 76 and 91 weeks
Population: Modified intent-to-treat (mITT) population, which included all participants who had taken at least 1 dose of double-blind investigational product and had at least 1 post-randomization DAS28 evaluation.
Measure: Number; unit: Participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Participants | 40 | 26 | 15
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — The rate of sustained remission was analyzed using a logistic regression model with a 2-sided significance level of 5%; Values are based on a logistic regression model with treatment as the only factor; Odds Ratio (OR) = 5.8, 95% CI 2-sided [2.7 to 12.5]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0085, Regression, Logistic — The rate of sustained remission was analyzed using a logistic regression model with a 2-sided significance level of 5%; Values are based on a logistic regression model with treatment as the only factor; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.3 to 5.3]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0397, Regression, Linear — The rate of sustained remission was analyzed using a logistic regression model with a 2-sided significance level of 5%; Values are based on a logistic regression model with treatment as the only factor; Odds Ratio (OR) = 2.22, 95% CI 2-sided [1.0 to 4.8]

2. Secondary Outcome: Number of Participants Achieving Complete Response (Using Disease Activity Score Based on 28-joint Count, Modified Total Sharp Score, Health Assessment Questionnaire)
Description: The composite measure of complete response over the last 3 months of Phase 1 was defined as:
  1. DAS28 <2.6 at the week 39 and 52 visits and,
  2. No radiographic progression during Phase 1, defined as mean change in modified total Sharp score (mTSS) ≤0.5 and,
  3. Health Assessment Questionnaire (HAQ) ≤ 0.5 at the week 39 and week 52 visits
Time Frame: End of Phase 1
Population: Efficacy data were analyzed in the modified intent-to-treat (mITT) population, which included all participants who took at least 1 dose of open-label investigational product
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants | 89
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Binomial test-value tests the null hypothesis that the proportion is significantly different from 0. End of Phase 1; Test type: Superiority or Other; p < 0.0001, Binomial test

3. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 52 and Final on Therapy
Description: mTSS = sum of erosion and Joint Space Narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change: scores at observation minus score at baseline. An increase in mTSS from baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: 52 week and Final on Therapy (includes all visits for a participant up to Week 52 or the visit they discontinued at)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Units on a scale
  Week 52 (N = 200) | 0.3 (3.0)
  Final on Therapy (N = 269) | 0.4 (2.8)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 52; Test type: Superiority or Other; p = 0.1183, Paired t-test
Statistical Analysis 2: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Final on therapy; Test type: Superiority or Other; p = 0.0286, Paired t-test

4. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire: Percent Overall Work Impairment Due to Problem
Description: WPAI:6 question participant rated questionnaire to determine the degree to which rheumatoid arthritis affected work productivity while at work and affected activities outside of work. Four scores are derived:percentage of absenteeism, percentage of presenteeism (reduced productivity while at work),overall work impairment score that combined absenteeism and presenteeism and percentage of impairment in activities performed outside of work. Scores scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher scores indicated greater impairment and less productivity. The raw scores (0-10) are converted to percents (the variable is named "Percent impairment While Working") and as such range from 0 to 100.
Time Frame: 13, 26, 39, 52 weeks and Final on Therapy (includes all visits for a participant up to Week 52 or the visit they discontinued at)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
units on a scale
  Week 13 (N = 100) | -27.6 (27.4)
  Week 26 (N = 94) | -32.2 (28.0)
  Week 39 (N = 97) | -35.9 (27.0)
  Week 52 (N = 81) | -37.3 (30.7)
  Final on Therapy (N = 124) | -35.5 (31.3)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 13, 26, 39, 52 and final on therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test

5. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire: Percent Impairment While Working Due to Problem
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
units on a scale
  Week 13 (N = 140) | -27.1 (27.8)
  Week 26 (N = 138) | -31.5 (28.0)
  Week 39 (N = 129) | -35.3 (27.3)
  Week 52 (N = 116) | -36.6 (31.5)
  Final on Therapy (N = 169) | -33.7 (30.3)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 13, 26, 39, 52 and final on therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test

6. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire: Percent Work Time Missed Due to Problem
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
units on a scale
  Week 13 (N = 116) | -8.9 (34.5)
  Week 26 (N = 110) | -8.8 (32.5)
  Week 39 (N = 110) | -9.0 (30.7)
  Week 52 (N = 93) | -12.9 (32.4)
  Final on Therapy (N = 138) | -10.7 (35.3)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 13; Test type: Superiority or Other; p = 0.0063, Paired t-test
Statistical Analysis 2: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 26; Test type: Superiority or Other; p = 0.0053, Paired t-test
Statistical Analysis 3: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 39; Test type: Superiority or Other; p = 0.0027, Paired t-test
Statistical Analysis 4: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 52; Test type: Superiority or Other; p = 0.0002, Paired t-test
Statistical Analysis 5: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Final on therapy; Test type: Superiority or Other; p = 0.0005, Paired t-test

7. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire: Percent Activity Impairment Due to Problem
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
units on a scale
  Week 13 (N = 244) | -30.3 (26.0)
  Week 26 (N = 241) | -34.7 (27.5)
  Week 39 (N = 224) | -39.9 (27.0)
  Week 52 (N = 194) | -41.3 (28.6)
  Final on Therapy (N = 270) | -36.4 (29.4)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 13, 26, 39, 52 and final on therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test

8. Secondary Outcome: Number of Participants Achieving American College of Rhematology 20% (ACR 20) Response
Description: ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: 2, 4, 8, 13, 26, 39, 52 weeks and Final on Therapy (includes all visits for a participant up to Week 52 or the visit they discontinued at)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants
  Week 2 (N = 297) | 139
  Week 4 (N = 295) | 195
  Week 8 (N = 290) | 225
  Week 13 (N = 280) | 232
  Week 26 (N = 272) | 232
  Week 39 (N = 256) | 235
  Week 52 (N = 221) | 212
  Final on Therapy (N = 301) | 258
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Binomial test-value tests the null hypothesis that the proportion is significantly different from 0. Week 2, 4, 8, 13, 26, 39, 52 and final on therapy; Test type: Superiority or Other; p < 0.0001, Binomial test

9. Secondary Outcome: Number of Participants Achieving American College of Rhematology 50% (ACR 50) Response
Description: ACR50 response: greater than or equal to (≥) 50 percent (%) improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants
  Week 2 (N = 297) | 52
  Week 4 (N = 295) | 114
  Week 8 (N = 290) | 144
  Week 13 (N = 280) | 169
  Week 26 (N = 272) | 190
  Week 39 (N = 256) | 218
  Week 52 (N = 221) | 202
  Final on Therapy (N = 301) | 229
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Binomial test-value tests the null hypothesis that the proportion is significantly different from 0. Week 2, 4, 8, 13, 26, 39, 52 week and final on therapy; Test type: Superiority or Other; p < 0.0001, Binomial test

10. Secondary Outcome: Number of Participants Achieving American College of Rhematology 70% (ACR 70) Response
Description: ACR70 response: greater than or equal to (≥) 70 percent (%) improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants
  Week 2 (N = 297) | 17
  Week 4 (N = 295) | 49
  Week 8 (N = 290) | 80
  Week 13 (N = 280) | 115
  Week 26 (N = 272) | 146
  Week 39 (N = 256) | 178
  Week 52 (N = 221) | 176
  Final on Therapy (N = 301) | 198
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test

11. Secondary Outcome: Number of Participants Achieving American College of Rhematology 90% (ACR 90) Response
Description: ACR90 response: greater than or equal to (≥) 90 percent (%) improvement in tender or swollen joint counts and 90% improvement in 3 of the following 5 criteria: 1) physician's global assessment of disease activity, 2) subject's assessment of disease activity, 3) subject's assessment of pain, 4) subject's assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants
  Week 2 (N = 297) | 2
  Week 4 (N = 295) | 11
  Week 8 (N = 290) | 22
  Week 13 (N = 280) | 34
  Week 26 (N = 272) | 70
  Week 39 (N = 256) | 85
  Week 52 (N = 221) | 97
  Final on Therapy (N = 301) | 105
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test

12. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 100 Visual Analog Scale (VAS), with 0 = no disease activity and 100 = extreme disease activity.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Units on a scale
  Week 2 (N = 300) | -21.1 (18.2)
  Week 4 (N = 299) | -29.9 (19.7)
  Week 8 (N = 294) | -34.8 (19.9)
  Week 13 (N = 284) | -38.7 (20.0)
  Week 26 (N = 277) | -42.4 (18.9)
  Week 39 (N = 260) | -46.5 (18.5)
  Week 52 (N = 223) | -49.2 (17.2)
  Final on Therapy (N = 305) | -45.0 (19.8)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 2, 4, 8, 13, 26, 39, 52 week and final on therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test

13. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity
Description: Participant's Global Assessment of Disease Activity was measured on a 0 to 100 mm Visual Analog Scale (VAS), with 0 mm = no disease activity and 100 = extreme disease activity
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
units on a scale
  Week 2 (N = 301) | -23.4 (24.4)
  Week 4 (N = 299) | -27.4 (26.2)
  Week 8 (N = 294) | -31.8 (26.0)
  Week 13 (N = 285) | -34.6 (26.8)
  Week 26 (N = 277) | -40.1 (28.1)
  Week 39 (N = 260) | -44.8 (26.6)
  Week 52 (N = 233) | -48.6 (26.2)
  Final on Therapy (N = 305) | -42.8 (28.4)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); Significance tests were based on paired t-tests using a 2-sided α=0.05. Week 2, 4, 8, 13, 26, 39, 52 and final on therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test

14. Secondary Outcome: Change From Baseline in DAS44 Score at All Visits
Description: DAS44 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 44 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS44 <1.6 = clinical remission, DAS44 ≤2.4 = low disease activity.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
units on a scale
  Week 2 (N = 297) | -1.3 (0.9)
  Week 4 (N = 293) | -1.9 (1.1)
  Week 8 (N = 293) | -2.3 (1.1)
  Week 13 (N = 282) | -2.5 (1.2)
  Week 26 (N = 276) | -2.9 (1.2)
  Week 39 (N = 259) | -3.2 (1.2)
  Week 52 (N = 221) | -3.4 (1.2)
  Final on Therapy (N = 305) | -3.0 (1.3)
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p < 0.0001, Paired t-test

15. Secondary Outcome: Number of Participants With Disease Activity Score Based on 44-joints Count (DAS44)-Remission
Description: as for outcome 14
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants
  Week 2 (N = 297) | 13
  Week 4 (N = 293) | 48
  Week 8 (N = 293) | 81
  Week 13 (N = 282) | 95
  Week 26 (N = 276) | 142
  Week 39 (N = 259) | 174
  Week 52 (N = 221) | 193
  Final on Therapy (N = 305) | 211
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test

16. Secondary Outcome: Number of Participants With Disease Activity Score Based on 44-joints Count (DAS44) - Low Disease Activity
Description: as for outcome 14
Time Frame: as for outcome 8
Population: Efficacy data were analyzed in the modified intent-to-treat (mITT) population, which included all participant who took at least 1 dose of open-label investigational product
Measure: Number; unit: participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
participants
  Week 2 (N = 297) | 67
  Week 4 (N = 293) | 122
  Week 8 (N = 293) | 157
  Week 13 (N = 282) | 194
  Week 26 (N = 276) | 210
  Week 39 (N = 259) | 236
  Week 52 (N = 221) | 214
  Final on Therapy (N = 305) | 249
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Binomial test

17. Secondary Outcome: Proportion of Subjects Achieving a Patient Acceptable Symptom State (PASS) at Each Visit
Description: The PASS is defined as a symptom state that the participants consider acceptable.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | ETN 50 QW + MTX (Phase 1)
Number analyzed (Participants) | 306
Participants
  Week 2 (N = 297) | 151
  Week 4 (N = 292) | 180
  Week 8 (N = 288) | 189
  Week 13 (N = 279) | 197
  Week 26 (N = 268) | 213
  Week 39 (N = 257) | 219
  Week 52 (N = 220) | 206
  Final on Therapy (N = 305) | 250
Statistical Analysis 1: Comparison: ETN 50 QW + MTX (Phase 1); P-value is from McNemar's test for no change from baseline in response rate. Week 2, 4, 8, 13, 26, 39, 52 week and final on therapy; Test type: Superiority or Other; p < 0.0001, McNemar

18. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: 52, 56, 64, 76, 91 weeks and Final on Therapy (includes all visits for a participant up to Week 91 or the visit they discontinued at)
Population: Modified intent-to-treat (mITT) population, which included all subjects who had taken at least 1 dose of double-blind investigational product and had at least 1 post-randomization DAS28 evaluation.
Measure: Number; unit: participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
participants
  Week 52 (N = 63, 63, 65) | 61 | 63 | 64
  Week 56 (N = 63, 63, 63) | 59 | 59 | 56
  Week 64 (N = 62, 61, 62) | 61 | 51 | 44
  Week 76 (N = 60, 55, 46) | 57 | 51 | 40
  Week 91 (N = 57, 50, 38) | 55 | 48 | 31
  Final on Therapy (N = 63, 63, 65) | 58 | 52 | 37
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.4075, Longitudinal statistical model; Odds ratios and p-values are based on a longitudinal statistical model with factors for treatment, visit, and interaction of treatment and visit; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.4 to 7.6]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0011, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 8.88, 95% CI 2-sided [2.4 to 33.1]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0031, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 4.87, 95% CI 2-sided [1.7 to 13.9]

19. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: as for outcome 9
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
participants
  Week 52 (N = 63, 63, 65) | 58 | 61 | 62
  Week 56 (N = 63, 63, 63) | 55 | 58 | 48
  Week 64 (N = 62, 61, 62) | 59 | 47 | 33
  Week 76 (N = 60, 55, 46) | 54 | 48 | 33
  Week 91 (N = 57, 50, 38) | 48 | 45 | 29
  Final on Therapy (N = 63, 63, 65) | 50 | 47 | 32
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.5951, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.3 to 2.0]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0934, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.9 to 5.5]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0314, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 2.85, 95% CI 2-sided [1.1 to 7.4]

20. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: as for outcome 10
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
participants
  Week 52 (N = 63, 63, 65) | 52 | 56 | 52
  Week 56 (N = 63, 63, 63) | 46 | 51 | 37
  Week 64 (N = 62, 61, 62) | 49 | 42 | 24
  Week 76 (N = 60, 55, 46) | 47 | 41 | 25
  Week 91 (N = 57, 50, 38) | 44 | 39 | 25
  Final on Therapy (N = 63, 63, 65) | 46 | 39 | 26
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.6152, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.5 to 2.8]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0432, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.0 to 5.4]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.1189, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.8 to 4.3]

21. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 90% (ACR90) Response
Description: as for outcome 11
Time Frame: 52, 64, 76, 91 weeks and Final on Therapy (includes all visits for a participant up to Week 91 or the visit they discontinued at)
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
participants
  Week 52 (N = 63, 63, 65) | 32 | 31 | 25
  Week 56 (N = 63, 63, 63) | 32 | 31 | 20
  Week 64 (N = 62, 61, 62) | 29 | 22 | 11
  Week 76 (N = 60, 55, 46) | 25 | 18 | 13
  Week 91 (N = 57, 50, 38) | 30 | 19 | 12
  Final on Therapy (N = 63, 63, 65) | 31 | 19 | 12
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0535, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.0 to 4.7]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0064, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.4 to 7.5]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.3696, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.6 to 3.6]

22. Secondary Outcome: Number of Participants With Disease Activity Score Based on 44-joints Count (DAS44) Remission
Description: as for outcome 14
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Participants
  Week 52 (N = 63, 65, 65) | 60 | 62 | 60
  Week 56 (N = 63, 65, 63) | 52 | 52 | 47
  Week 64 (N = 62, 63, 60) | 54 | 44 | 25
  Week 76 (N = 60, 57, 46) | 51 | 42 | 24
  Week 91 (N = 57, 52, 38) | 48 | 39 | 23
  Final on Therapy (N = 63, 65, 65) | 51 | 40 | 24
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0788, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.9 to 5.2]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0007, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 4.57, 95% CI 2-sided [1.9 to 11.0]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0676, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.9 to 4.7]

23. Secondary Outcome: Number of Participants With Disease Activity Score Based on 44-joints Count (DAS44) - Low Disease Activity
Description: as for outcome 14
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Participants
  Week 52 (N = 63, 65, 65) | 63 | 65 | 65
  Week 56 (N = 63, 65, 63) | 62 | 60 | 54
  Week 64 (N = 62, 63, 60) | 61 | 52 | 38
  Week 76 (N = 60, 57, 46) | 57 | 54 | 37
  Week 91 (N = 57, 52, 38) | 56 | 47 | 33
  Final on Therapy (N = 63, 65, 65) | 60 | 50 | 35
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0548, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 7.56, 95% CI 2-sided [1.0 to 59.5]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0166, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 12.18, 95% CI 2-sided [1.6 to 94.2]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.3619, Longitudinal statistical model; [statistical method as in outcome 18, analysis 1]; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.6 to 4.5]

24. Secondary Outcome: Number of Participants Achieving Complete Response (Using Disease Activity Score Based on a 28-joint Count, Modified Total Sharp Score, Health Assessment Questionnaire)
Description: The composite measure of complete response over the last 3 months of Phase 2 was defined as:
  1. DAS28 <2.6 at the Week 76 and Week 91 visits and
  2. No radiographic progression during Phase 2, defined as mean change from Week 52 in mTSS of ≤0.5.
  3. Participant must achieve HAQ score ≤0.5 at Week 76 and 91 visits. HAQ is self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ score range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation.A subject had to satisfy all 3 criteria at thevisits to be defined as a responder
Time Frame: 52 and 91 weeks
Population: as for outcome 18
Measure: Number; unit: Participants
Groups:
- MTX + PBO (Phase 2): In Phase 2 MTX + PBO arm, the weekly dose of etanercept was tapered from the 50 mg dosage. At Week 52, subjects assigned to this arm received a double blinded 25 mg dose of etanercept as a subcutaneous injection using a pre filled syringe. All weekly doses thereafter (ie, Weeks 53 to 90) were administered as an etanercept matching placebo injection using a pre-filled syringe.Methotrexate was administered once weekly as oral capsules. All subjects received a dose of methotrexate during this Phase 2 study that was equal to their optimal methotrexate dose in earlier Phase 1 study.The subjects received the study treatment for 39 weeks, unless the subject was evaluated as non-responder at Week 64 or Week 76 and discontinued the study. Participants in sustained remission (Disease Activity Score based on 28-joints count [DAS28] <2.6) or with low disease activity (2.6 = DAS28 = 3.2) at Week 91 were classified as Phase 2 responder, and will continue to Phase 3 study
- Placebo (PBO) (Phase 2): In Phase 2 Placebo (PBO) arm, the weekly dose of etanercept was tapered from the 50 mg dosage to a placebo injection. At Week 52, subjects assigned to this arm received a double blinded 25 mg dose of etanercept as a subcutaneous injection using a pre filled syringe.All weekly doses thereafter (ie, Weeks 53 to 90) were administered as an etanercept-matching placebo injection using a pre-filled syringe.Methotrexate-matching placebo was administered once weekly as oral capsules. The subjects received the study treatment for 39 weeks, unless the subject was evaluated as non-responder at Week 64 or Week 76 and discontinued the study. Participants in sustained remission (Disease Activity Score based on 28-joints count [DAS28] <2.6) or with low disease activity (2.6 = DAS28 = 3.2) at Week 91 were classified as Phase 2 responder, and will continue to Phase 3 study
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Participants | 36 | 19 | 7
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0017, Regression, Logistic; Odds ratios, p-values, and 95% CIs are based on a logistic regression model with treatment as the only factor; Odds Ratio (OR) = 3.23, 95% CI 2-sided [1.6 to 6.7]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds ratios, p-values, and 95% CIs are based on a logistic regression model with treatment as the only factor; Odds Ratio (OR) = 11.05, 95% CI 2-sided [4.4 to 28.0]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0111, Regression, Logistic; Odds ratios, p-values, and 95% CIs are based on a logistic regression model with treatment as the only factor; Odds Ratio (OR) = 3.42, 95% CI 2-sided [1.3 to 8.8]

25. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: as for outcome 12
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 52 (N = 63, 65, 65) | 5.0 (5.3) | 4.2 (4.9) | 6.3 (8.0)
  Week 56 (N = 63, 65, 65) | 5.5 (6.2) | 7.7 (12.6) | 12.2 (15.1)
  Week 64 (N = 62, 63, 62) | 6.0 (7.4) | 11.6 (16.7) | 23.6 (26.0)
  Week 76 (N = 60, 57, 46) | 5.5 (7.1) | 9.0 (13.6) | 14.6 (18.1)
  Week 91 (N = 57, 52, 38) | 5.8 (9.8) | 10.3 (16.8) | 15.9 (21.7)
  Final on Therapy (N = 63, 65, 65) | 6.9 (10.8) | 16.7 (21.7) | 30.7 (28.4)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0328, Longitudinal statistical model; Values are based on a longitudinal statistical model with factors for Week 52 value, treatment, visit, and interaction of treatment; Mean Difference (Final Values) = -8.66, 95% CI 2-sided [-16.6 to -0.7]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p < 0.0001, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -21.64, 95% CI 2-sided [-30.1 to -13.2]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0035, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -12.98, 95% CI 2-sided [-21.5 to -4.5]

26. Secondary Outcome: Participant's Global Assessment of Disease Activity
Description: as for outcome 13
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 52 (N = 63, 65, 65) | 5.8 (6.3) | 5.7 (7.7) | 9.3 (14.1)
  Week 56 (N = 63, 65, 65) | 10.3 (14.8) | 9.7 (16.3) | 17.3 (22.1)
  Week 64 (N = 62, 63, 62) | 7.6 (9.1) | 17.8 (25.5) | 31.0 (31.4)
  Week 76 (N = 60, 56, 46) | 8.9 (12.1) | 11.7 (17.9) | 18.3 (18.7)
  Week 91 (N = 56, 52, 38) | 9.6 (14.1) | 12.3 (17.5) | 18.8 (25.7)
  Final on Therapy (N = 63, 65, 65) | 11.1 (16.2) | 20.7 (25.9) | 37.1 (33.9)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.2473, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -4.36, 95% CI 2-sided [-11.8 to 3.1]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0016, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -13.19, 95% CI 2-sided [-21.3 to -5.1]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0348, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -8.83, 95% CI 2-sided [-17.0 to -0.6]

27. Secondary Outcome: Participant's Global Assessment of Pain (Visual Analogue Scale) (VAS)
Description: 100-mm line (Visual Analog Scale) marked by the participant to measure their degree of pain over past 2-3 weeks. Range: 0 = no pain to 100 = pain as bad as it could be.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
mm
  Week 52 (N = 63, 65, 65) | 7.3 (7.7) | 6.9 (8.6) | 9.9 (14.8)
  Week 56 (N = 63, 65, 65) | 10.9 (15.0) | 10.2 (16.9) | 18.8 (23.1)
  Week 64 (N = 62, 63, 62) | 8.0 (9.8) | 18.0 (25.1) | 31.7 (31.3)
  Week 76 (N = 60, 56, 46) | 9.8 (12.9) | 12.3 (19.2) | 17.6 (18.1)
  Week 91 (N = 57, 52, 38) | 9.5 (12.7) | 13.3 (16.4) | 19.7 (26.1)
  Final on Therapy (N = 63, 65, 65) | 11.4 (15.4) | 21.4 (24.8) | 37.8 (33.7)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.1248, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -5.51, 95% CI 2-sided [-12.6 to 1.6]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0004, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -14.14, 95% CI 2-sided [-21.8 to -6.5]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0306, Longitudinal statistical model; [statistical method as in outcome 25, analysis 1]; Mean Difference (Final Values) = -8.63, 95% CI 2-sided [-16.4 to -0.8]

28. Secondary Outcome: Number of Participants Achieving Patient Acceptable Symptom State (PASS)
Description: The PASS is defined as a symptom state that the subjects consider acceptable.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Participants
  Week 52 (N = 61, 65, 64) | 57 | 64 | 61
  Week 56 (N = 63, 63, 64) | 57 | 58 | 53
  Week 64 (N = 61, 60, 60) | 58 | 51 | 42
  Week 76 (N = 60, 56, 45) | 57 | 48 | 38
  Week 91 (N = 57, 52, 38) | 52 | 46 | 33
  Final on Therapy (N = 63, 65, 65) | 56 | 50 | 38
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.4717, Longitudinal statistical model; Values are based on a longitudinal statistical model with factors for treatment, visit, and interaction of treatment and visit; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.5 to 4.6]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0551, Longitudinal statistical model; [statistical method as in outcome 28, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.0 to 7.8]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.2141, Longitudinal statistical model; [statistical method as in outcome 28, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.7 to 4.8]

29. Secondary Outcome: Modified Total Sharp Score (mTSS) at Week 52
Description: mTSS = sum of erosion and Joint Space Narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change: scores at observation minus score at baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: 52 weeks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 58 | 56 | 49
Units on a scale | 8.4 (13.5) | 8.4 (15.1) | 8.6 (12.8)

30. Secondary Outcome: Change From Baseline mTSS at Week 91 and Final on Therapy
Description: as for outcome 29
Time Frame: 91 weeks and Final on Therapy (includes all visits for a participant up to Week 91 or the visit they discontinued at)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 91 (N = 51, 45, 30) | 0.0 (0.16) | 0.0 (0.17) | 0.5 (0.21)
  Final on Therapy (N = 58, 56, 49) | 0.1 (0.14) | -0.0 (0.15) | 0.4 (0.16)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.9652, ANCOVA; P-values for between-treatment comparisons are based on ANCOVA on ranks of change in score with ranks of Week 52 value as covariate; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.5 to 0.4]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.2168, ANCOVA; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.0 to 0.0]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.2131, ANCOVA; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.0 to 0.0]

31. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire: Percent Work Time Missed in the Past 7 Days Due to Problem
Description: WPAI: 6 question participant rated questionnaire to determine the degree to which rheumatoid arthritis affected work productivity while at work and affected activities outside of work. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combined absenteeism and presenteeism and percentage of impairment in activities performed outside of work. Scores scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher scores indicated greater impairment and less productivity. The raw (0-10) scores are converted to percents (the variable is named "Percent impairment While Working") and as such range from 0 to 100.
Time Frame: 52 weeks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 29 | 43 | 25
units on a scale | 0.2 (1.2) | 0.1 (0.6) | 0.0 (0.0)

32. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Percent Work Time Missed in the Past 7 Days Due to Problem
Description: WPAI is a 6 question participant rated questionnaire determined the degree to which rheumatoid arthritis affected work productivity while at work and affected activities outside of work. Scores scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher scores = greater impairment and less productivity. The raw (0-10) scores were converted to percent (the variable is named "Percent impairment While Working") and as such range from 0 to 100.
Time Frame: 64, 76, 91 weeks and Final on Therapy (includes all visits for a participant upto Week 91 or the visit they discontinued at)
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 64 (N = 30, 44, 26) | 1.9 (2.78) | 2.6 (2.29) | 6.1 (3.04)
  Week 76 (N = 28, 33, 18) | -0.1 (2.38) | 2.9 (2.19) | 2.6 (3.09)
  Week 91 (N = 29, 32, 14) | 4.4 (3.78) | 4.0 (3.63) | 7.0 (5.79)
  Final on Therapy (N = 34, 48, 29) | 3.6 (3.65) | 5.3 (3.07) | 10.2 (4.06)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hyothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.9338, ANCOVA; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-10.0 to 10.9] — Values are based on a model with factors for Week 52 value, treatment, visit, and interaction of treatment and Week 52 value and treatment and visit
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.7130, ANCOVA; Values are based on a model with factors for Week 52 value, treatment, visit, and interaction of treatment and Week 52 value and treatment and visit; Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-16.4 to 11.2]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.6628, ANCOVA; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-16.6 to 10.6]

33. Secondary Outcome: WPAI Questionnaire: Percent Impairment While Working in the Past 7 Days Due to Problem
Description: as for outcome 31
Time Frame: 52 Weeks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
units on a scale | 6.2 (9.2) | 8.9 (15.5) | 14.2 (17.9)

34. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Percent Impairment While Working in the Past 7 Days Due to Problem
Description: WPAI: 6 question participant rated questionnaire determined the degree to which rheumatoid arthritis affected work productivity while at work and affected activities outside of work. Scores scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher scores = greater impairment and less productivity. The raw (0-10) scores were converted to percent (the variable is named "Percent impairment While Working") and as such range from 0 to 100.
Time Frame: as for outcome 32
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 64 (N = 37, 49, 31) | -2.5 (3.57) | 9.6 (3.16) | 18.2 (3.96)
  Week 76 (N = 38, 38, 23) | -0.6 (2.16) | 2.3 (2.01) | 12.2 (2.54)
  Week 91 (N = 37, 35, 18) | 1.8 (3.16) | 8.6 (3.06) | 18.4 (4.23)
  Final on Therapy (N = 45, 50, 40) | 1.1 (3.51) | 11.1 (3.10) | 19.9 (3.76)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.1303, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -6.74, 95% CI 2-sided [-15.5 to 2.0]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0024, Longitudinal statisitical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -16.59, 95% CI 2-sided [-27.1 to -6.0]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0621, Longitudinal statistical model; Mean Difference (Final Values) = -9.85, 95% CI 2-sided [-20.2 to 0.5]

35. Secondary Outcome: WPAI Questionnaire: Percent Overall Work Impairment in the Past 7 Days Due to Problem
Description: as for outcome 31
Time Frame: 52 weeks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 27 | 42 | 24
units on a scale | 5.3 (9.8) | 6.7 (15.0) | 9.2 (12.8)

36. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Percent Overall Work Impairment in the Past 7 Days Due to Problem
Description: as for outcome 34
Time Frame: as for outcome 32
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 64 (N = 29, 43, 25) | 0.1 (4.49) | 11.5 (3.75) | 22.4 (2.01)
  Week 76 (N = 27, 30, 18) | -0.9 (2.40) | 2.6 (2.18) | 16.6 (2.95)
  Week 91 (N = 28, 30, 13) | 5.4 (3.98) | 9.5 (3.74) | 22.0 (5.75)
  Final on Therapy (N = 34, 48, 28) | 4.4 (4.32) | 13.3 (3.60) | 25.1 (4.84)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.4664, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -4.01, 95% CI 2-sided [-15.0 to 6.9]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0210, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -16.57, 95% CI 2-sided [-30.6 to -2.6]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0713, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -12.56, 95% CI 2-sided [-26.2 to 1.1]

37. Secondary Outcome: WPAI Questionnaire: Percent Activity Impairment in the Past 7 Days Due to Problem
Description: as for outcome 31
Time Frame: 52 weeks
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 56 | 60 | 60
Units on a scale | 8.6 (11.0) | 10.0 (15.9) | 16.8 (20.0)

38. Secondary Outcome: Change From Baseline in WPAI Questionnaire: Percent Activity Impairment in the Past 7 Days Due to Problem
Description: as for outcome 34
Time Frame: as for outcome 32
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2)
Number analyzed (Participants) | 63 | 65 | 65
Units on a scale
  Week 64 (N = 56, 60, 57) | -0.5 (3.21) | 9.9 (3.10) | 19.1 (3.18)
  Week 76 (N = 57, 55, 41) | 2.9 (2.94) | 7.1 (2.96) | 13.9 (3.35)
  Week 91 (N = 53, 49, 37) | -1.8 (2.83) | 7.3 (2.87) | 17.9 (3.20)
  Final on Therapy (N = 60, 64, 64) | -0.9 (3.24) | 12.2 (3.13) | 24.2 (3.16)
Statistical Analysis 1: Comparison: E25 + MTX (Phase 2) vs MTX + PBO (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0256, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -9.11, 95% CI 2-sided [-17.1 to -1.1]
Statistical Analysis 2: Comparison: E25 + MTX (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p < 0.0001, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -19.62, 95% CI 2-sided [-28.1 to -11.1]
Statistical Analysis 3: Comparison: MTX + PBO (Phase 2) vs Placebo (PBO) (Phase 2); Change from Week 52 to Week 91. The hypothesis of primary interest was the superiority of E25+MTX compared with PBO; Test type: Superiority or Other; p = 0.0161, Longitudinal statistical model; [statistical method as in outcome 32, analysis 2]; Mean Difference (Final Values) = -10.51, 95% CI 2-sided [-19.0 to -2.0]

ADVERSE EVENTS:
Time Frame: Screening to Week 117 (Phase 1, 2, and 3 data)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | ETN 50 QW + MTX (Phase 1) | E25 + MTX (Phase 2) | MTX + PBO (Phase 2) | Placebo (PBO) (Phase 2) | E25+MTX (Phase 3) | MTX (Phase 3) | Placebo (PBO) (Phase 3)
Serious Adverse Events (participants affected / at risk) | 28/306 | 3/63 | 2/65 | 2/65 | 0/53 | 0/46 | 2/32
Other Adverse Events (participants affected / at risk) | 130/306 | 10/63 | 8/65 | 11/65 | 13/53 | 8/46 | 4/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETN 50 QW + MTX (Phase 1) (N=306) | E25 + MTX (Phase 2) (N=63) | MTX + PBO (Phase 2) (N=65) | Placebo (PBO) (Phase 2) (N=65) | E25+MTX (Phase 3) (N=53) | MTX (Phase 3) (N=46) | Placebo (PBO) (Phase 3) (N=32)
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear canal stenosis postoperative (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis Erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infected Cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Systemic Sclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss Of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric Decompensation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETN 50 QW + MTX (Phase 1) (N=306) | E25 + MTX (Phase 2) (N=63) | MTX + PBO (Phase 2) (N=65) | Placebo (PBO) (Phase 2) (N=65) | E25+MTX (Phase 3) (N=53) | MTX (Phase 3) (N=46) | Placebo (PBO) (Phase 3) (N=32)
Nausea (Gastrointestinal disorders) | 39 | 0 | 0 | 0 (0) | 0 | 0 | 0
Injection site Erythema (General disorders) | 17 | 0 | 0 | 0 (0) | 0 | 0 | 0
Injection site reaction (General disorders) | 19 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 39 | 5 | 3 | 3 | 3 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 4 | 3 | 3 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 17 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 20 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 6 | 10 | 7 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.